CLINICAL TRIAL: NCT00463658
Title: The Comparative Effects and Expenses of a Proactive Nurse-Led, Multifactorial and Interdisciplinary Team Approach to Falls Prevention for Older At-Risk Home Care Clients
Brief Title: Interdisciplinary Falls Prevention for Seniors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Patient Safety Institute (Other); Mississauga Halton Community Care Access Centre (Unknown); Hamilton Niagara Haldimand Brant Community Care Access Centre (Other); Ontario Ministry of Health and Long Term Care (Other Government); Halton Region Health Department (Other); Community Rehab (Unknown)
Responsible Party: Ms. Marie Townsend, Committee on Scientific Development, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RFAAA0506164
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Injuries
Keywords: Falls; Home Care; Aging Population; Clinical Effectiveness; Health Economics
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects in the interdisciplinary group received home care services from a team of professional service providers (CCAC Case Manager, Registered Nurse, Occupational Therapist, Physiotherapist, Registered Dietician) with experience and training in falls prevention. The team provided a comprehensive, coordinated and evidence based approach to falls prevention through regular home visits, weekly case conferencing, a single accessible fall prevention plan,and joint client visits.
  Interventions: Other: Falls Prevention
- 2 (No Intervention): Participants allocated to the control group received standard home care services arranged by the CCAC. These include routine follow-up by the CCAC case manager whose focus is on assessing client's eligibility for in-home health services, arrangement and coordination of professional (i.e. nursing, occupational therapy, physiotherapy, social work, speech-language pathology, nutrition) and non-professional HSS, information and referral to community agencies, and ongoing monitoring and evaluating the plan of care through in-home assessments with clients.

INTERVENTIONS:
Other: Falls Prevention — Subjects in the interdisciplinary group will receive home care services from a team of professional service providers (CCAC Case Manager, Public Health Nurse (Registered Nurse), Occupational Therapist, Physiotherapist, Nutritionist) with experience and training in falls prevention. The team will provide a comprehensive, coordinated and evidence based approach to falls prevention through weekly case conferencing, a written interdisciplinary care plan, and joint client visits.
  Other Names: Interdisciplinary Falls Prevention Team
  Arms: 1

SUMMARY:
With an aging population, an associated increase in the number of falls and fall injuries, there is a need to examine how health care services, such as home care, can best prevent falls among older people. This project will directly address this area by evaluating the effects and expense of an innovative approach to home care service delivery for older people at-risk for falls.

DETAILED DESCRIPTION:
Falls and fall injuries are common-potentially preventable-causes of mortality, morbidity, functional decline, and increased health-care use and cost among community-living seniors over 75 years of age.

The knowledge gained from this project will directly address the Canadian Patient Safety Institute's priority areas for research in the Applied Health Services Research Stream by evaluating an innovative approach to reducing adverse events in a community-based (home care) setting.

The project will also identify the prevalence, determinants and costs of falls and fall injuries among older people requiring home care services. The design will be a two-armed; single blind randomized controlled trial of 110 older people 75 years and over, at risk for falls receiving hom care in Ontario. Subjects will be randomly allocated to either usual home care (control) or the interdisciplinary team. In the interdisciplinary group, a team of professional home care service providers, with specialized training in falls prevention, will proactively provide a comprehensive, coordinated and evidence based approach to falls prevention. The results will inform policies and practice related to the allocation and delivery of home care services for falls prevention across Canada.

ELIGIBILITY:
Inclusion Criteria:

* Must be English speaking
* 75 years of age and over
* Newly referred to and eligible for personal support services
* Living at home in the community
* Identified as being at risk for falls

Exclusion Criteria:

* Refusal to give informed consent
* Unable to read/write English and a translator is not available

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Number of self-reported falls: Falls surveillance report | 10 minutes

SECONDARY OUTCOMES:
Health-Related Quality of Life and Function: SF-36 Health Survey | 15-20 minutes
Gait and Balance: Performance-Oriented Mobility Assessment | 10 minutes
Depression: Centre for Epidemiological Studies in Depression Scale | 5-10 minutes
Standardized Mini Mental State Examination | 20-25 minutes
Confidence in Performing Activities of Daily Living: Modified Falls Efficacy Scale | 5-10 minutes
Nutritional risk: Screen II Questionnaire | 10-15 minutes
Cost of Use of Health Services: Health and Social Services Utilization Questionnaire | 20 minutes
Caregiver burden: Caregiver Strain Index | 5-10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, RN MScN PhD, Principal Investigator — School of Nursing, McMaster University
Locations (1):
- McMaster University - Faculty of Health Sciences at Frid, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Isaranuwatchai W, Perdrizet J, Markle-Reid M, Hoch JS. Cost-effectiveness analysis of a multifactorial fall prevention intervention in older home care clients at risk for falling. BMC Geriatr. 2017 Sep 1;17(1):199. doi: 10.1186/s12877-017-0599-9. PMID 28863774
- [Derived] Markle-Reid M, Browne G, Gafni A, Roberts J, Weir R, Thabane L, Miles M, Vaitonis V, Hecimovich C, Baxter P, Henderson S. The effects and costs of a multifactorial and interdisciplinary team approach to falls prevention for older home care clients 'at risk' for falling: a randomized controlled trial. Can J Aging. 2010 Mar;29(1):139-61. doi: 10.1017/S0714980809990377. PMID 20202271
- [Derived] Markle-Reid M, Browne G, Gafni A, Roberts J, Weir R, Thabane L, Miles M, Vaitonis V, Hecimovich C, Baxter P, Henderson S. A cross-sectional study of the prevalence, correlates, and costs of falls in older home care clients 'at risk' for falling. Can J Aging. 2010 Mar;29(1):119-37. doi: 10.1017/S0714980809990365. PMID 20202270